CLINICAL TRIAL: NCT05711706
Title: The Effect of Su Jok Application on Pain, Anxiety and Quality of Recovery After Lumbar Disc Surgery
Brief Title: Su Jok Application in After Lumbar Disc Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Niran Çoban (Other)
Responsible Party: Sponsor-Investigator, Niran Çoban, Lecturer, Doctor, Istanbul Gedik University
Organization: Istanbul Gedik University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: NC*
Record Dates: First submitted 2022-11-28; First posted 2023-02-03 (Actual); Last update posted 2024-03-26 (Actual); Status verified 2024-03

CONDITIONS: Pain, Postoperative; Lumbar Disc Herniation; Surgery; Nurse's Role
MeSH Terms: conditions — Pain, Postoperative; Intervertebral Disc Displacement

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Su Jok Application (Experimental): I. Interview: One Day Before Surgery:
  II. Interview: Post-Surgery - After Transfer to the Clinic III. Interview: Postoperative Day 1 IV. Interview: Postoperative Day 2 V. Interview (Post-Operative Day 10
  Interventions: Other: Su Jok Application
- Standard care (No Intervention): I. Interview: One Day Before Surgery:
  II. Interview: Post-Surgery - After Transfer to the Clinic III. Interview: Postoperative Day 1 IV. Interview: Postoperative Day 2 V. Interview (Post-Operative Day 10

INTERVENTIONS:
Other: Su Jok Application — Su Jok massage appplication
  Arms: Su Jok Application

SUMMARY:
Surgical treatment is applied in 15% of individuals diagnosed with lumbar disc herniation. In this study, it was aimed to determine the effect of Su Jok application, which is one of the non-drug methods, in reducing or completely eliminating pain and anxiety after lumbar disc surgery and increasing the quality of recovery.The universe of the study, between November 2022 and June 2023, Istanbul Kartal Dr. Patients with lumbar disc surgery will be recruited in the Neurosurgery Clinic of Lütfi Kırdar City Hospital. Data will be obtained with Introductory Information Form, McGill Pain Scale Short Form (SF-MPQ), Visual Analog Scale (Visual Comparison Scale) (VAS), STAII State Anxiety Scale, Quality of Recovery Questionnaire (QOR-40). The individual who will undergo lumbar disc surgery will be visited in the clinic one day before the surgery and will be informed about the study. The sampled individuals will be included in the intervention and control groups using a random number table created with MS Excel software. Su Jok will be applied to the patients included in the intervention group at the third hour after the operation. Before the application, Quality of Recovery Questionnaire (QOR-40), McGill Pain Scale Short Form and STAII State Anxiety Scale will be administered. After the application, the pain levels of the patients will be re-evaluated with the Visual Analogue Scale (Visual Comparison Scale) (VAS) and their anxiety levels will be re-evaluated with the STAII State Anxiety Scale. On the first and second days after the surgery, the patients will be visited again in the clinic and the Quality of Healing Questionnaire (QOR-40), Visual Analog Scale (Visual Comparison Scale) (VAS) and STAII State Anxiety Scales will be administered before the Su Jok application, and then the Su Jok application will be repeated.After the application, the pain levels of the patients will be re-evaluated with the Visual Analogue Scale (Visual Comparison Scale) (VAS) and their anxiety levels will be re-evaluated with the STAII State Anxiety Scale. Patients will be interviewed again at the control appointment 10 days after discharge, and their quality of recovery will be determined using the Quality of Healing Questionnaire (QOR-40). In the control group, pain, anxiety and healing quality levels will be determined in the same periods without any application.

DETAILED DESCRIPTION:
Chronic low back pain has become a common problem today and is seen as a phenomenon that directly affects the daily life of individuals and, in parallel, affects their psychological and socioeconomic status. There are many causes of back pain. The most common problem among these is Lumbar disc herniation (LDH). LDH, which causes low back pain, is a condition in which the nucleus pulposus degenerates the annulus and causes herniation and pain as a result of the deterioration of the structure of the lower lumbar vertebrae that carry the weight of the trunk. Surgical treatment is applied in 15% of individuals diagnosed with LDH. Postoperative nursing care is based on interventions for ensuring homeostasis, preventing the re-development of herniation, preventing complications and early diagnosis, and enabling the patient to perform daily life activities. Post-operative pain affects all systems, prolonging the patient's recovery period and prolonging their quality of life.In pain management, it is essential to try to control it with the aim of preventing and eliminating pain. In addition to being an effective method, pharmacological methods are also reported to be effective in non-pharmacological methods such as relaxation exercises, elimination of painful stimuli, position, touch, and speaking. The role of the nurse in controlling pain is quite large. For this reason, it is necessary to have high-level pain control knowledge by educating himself on non-pharmacological methods . One of the non-pharmacological methods is Su Jok, which is a massage technique. Su Jok is explained by the principle of the "fitness system", in which the hands and feet are a miniature replica of the body. There are tiny swellings called "ball conformity" on the reflection points of the hands and feet of the organ where the disease occurs.As a result of the pressure massage applied to the area where the swelling is located, pain and withdrawal sensation occur in the application area. This feeling shows that the right point for application has been determined . "Diagnostic probe" or "diagnostic stick" is used to determine the correct point.After the correct point is determined, these points are stimulated by using various applicators (rings, metal starlets, magnets, seeds, etc.) and appropriate plant seeds, and the energy flow is maintained. Massage with seeds are the most commonly used natural applicators for Su Jok massage application. Since seeds give life to plants, it is argued that there is a great energy inside them and this energy is a life-giving source that is in constant exchange with the external environment. The application is in the form of massaging the seeds suitable for the determined point on the hand and foot by fixing them with a plaster.The period of use of seeds can last from several hours to a day; For long-term use, daily seed change is required. It is ensured that the applied seed is massaged at certain intervals. Thanks to the door control mechanism, the pain sensation is eliminated with the applied seed massage. Since Su Jok application does not cause any side effects, it can be used in all age groups; The time to create a positive effect can vary from a few minutes to a few days. This application can be used in acute and chronic pain complaints.Although there are limited studies in the literature on Su Jok massage, Cruz and Munoz (2012) reported a decrease in pain frequency and severity as a result of the study conducted with patients with tension-type headache. Gonzales et al. (2011) applied Su Jok to patients with carpal tunnel syndrome and reported a reduction in pain and other symptoms as a result . In another study in which Su Jok massage was applied to cesarean section patients, it was found that the postoperative Su Jok application reduced the level of pain . There is no educational background required for the Su Jok massage application. Anyone who receives training can perform Su Jok massage . After receiving Su Jok training, each individual can manage their pain with this massage technique. When the literature is examined, it is seen that the studies on the application of Su Jok massage are limited. Especially the pain experienced in the post-operative period increases the anxiety level of individuals and affects the healing process. Therefore, it is aimed to eliminate the pain with the Su Jok massage application. In this study, it is aimed to determine the effect of Su Jok massage, which is one of the non-drug methods, in reducing or completely eliminating pain and anxiety after lumbar disc surgery and increasing the quality of recovery.

ELIGIBILITY:
Inclusion Criteria:

* • Having undergone lumbar disc surgery under general anesthesia

  * 18 years old and over,
  * At least 3 hours have passed from the analgesic administration,
  * Patients willing to participate in the study will be included in the study.

Exclusion Criteria:

* • Loss of sensation, amputation, injury, etc., which will prevent application in hands. the one which,

  * Patient-controlled analgesia (PCA) is applied,
  * Over 70 years old,
  * Using anxiolytic and sedative drugs,
  * Having a psychiatric illness,
  * Patients with communication barriers will not be included in the study. Exclusion Criteria
  * Those who lost their lives after the operation,
  * Unstable hemodynamic status,
  * Patients with a hospital stay of less than 72 hours (due to Su Jok application for 3 days) will be excluded from the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2023-03-10 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-08-30 (Actual)

PRIMARY OUTCOMES:
The Effect of Su Jok Application on Pain | 12 month
  Visual Analogue Scale:The Visual Analog Scale is a one-dimensional scale commonly used to measure pain intensity. VAS is a measuring tool with a length of 0-10 cm (0-100 mm).McGill Pain Scale Short Form (SF-MPQ):The scale will be used to determine the qualitative characteristics of pain in the initial pain assessment of patients. Since the aim of the study is to determine the effect of the non-pharmacological method used on existing pain, VAS will be used in the pain assessment before and after the application.Post-Surgery.After Transfer to the Clinic:Patients who have undergone lumbar disc surgery will be visited at the clinic for Su Jok application at the 3rd hour after surgery,Before the Su Jok application, the patient's pain status will be determined with the SF-MPQ15 minutes after the Su Jok application, the patient's pain status will be determined by the Visual Analogue Scale (VAS). These stages will be applied again on the 1st and 2nd days after the surgery.
The Effect of Su Jok Application on Anxiety | 12 month
  State Anxiety Inventory: In our study, the "State Anxiety Inventory" will be used before and after the procedure to evaluate the anxiety levels of the patients in a certain situation.The "State Anxiety Inventory (STAI-I)" is a tool that measures how the individual feels at a particular moment and situation, that is, the level of anxiety in that condition. Post-Surgery - After Transfer to the Clinic: Before the Su Jok application, the patient's anxiety status will be determined by the State-Trait Anxiety Inventory (STAI-I),For 30 minutes, the point where the seed is fixed will be massaged with the Su Jok technique,15 minutes after the Su Jok application, the patient's pain status will be determined by the State-Trait Anxiety Inventory (STAI-I).These stages will be applied again on the 1st and 2nd days after the surgery.
The Effect of Su Jok Application on Quality of Recovery | 12 month
  The Quality of Healing-40 Scale (QoR-40) consists of five sub-dimensions and 40 items. The sub-dimensions of the scale are emotional state, physical comfort, patient support, physical independence and pain. with the individual.Post-Surgery - After Transfer to the Clinic:Before the Su Jok application, the quality of recovery of the patient will be determined by the Quality of Healing-40 Scale (QoR-40), which covers 24 hours.
  These stages will be applied again on the 1st -2nd days after the surgery and Postoperative 10th Day.

CONTACTS AND LOCATIONS:
Overall Officials: Niran COBAN, Study Director — https://akademik.yok.gov.tr/AkademikArama/view/viewAuthor.jsp
Locations (1):
- Niran COBAN, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Özbayır, T. (2011). (in) Nörolojik Travmalar, Karadakovan, A. ve Eti Aslan, F. (Ed.), Dahili ve Cerrahi Hastalıklarda Bakım, Adana: Nobel Kitabevi, 2. Baskı: 1280-1284.
- [Background] Lurie JD, Tosteson TD, Tosteson AN, Zhao W, Morgan TS, Abdu WA, Herkowitz H, Weinstein JN. Surgical versus nonoperative treatment for lumbar disc herniation: eight-year results for the spine patient outcomes research trial. Spine (Phila Pa 1976). 2014 Jan 1;39(1):3-16. doi: 10.1097/BRS.0000000000000088. PMID 24153171
- [Background] Woo, PJ. Kendi Kendine Su Jok Doktor. İstanbul: Vesta Ofset Matbaacılık, 2010.
- [Background] Ivanov, P. (2018). Su Jok and Moxa. A Self-Trea a Self-Treatment Manual. Lavcıel, H.(edt). Bulgaria:MEDIKS Ltd
- [Background] Woo, J. W. (1987). Be Your Own Doctor. India: Smile Academy.
- [Background] Cruz, JC.P, Sotelo Matos, AM., Castaigne, YF., Pérez, AMP. Su-Jok Therapy for Cervicalgia Treatment. Correo Científico Médico de Holguín. 2018;4.
- [Background] Rodríguez, AC, Mendoza, YA, García, EFC, Castañeda YT. (2018). Su-Jok therapy in patients with cervicalgia diagnosis. Facultad de Tecnología de la Salud. 9(3):42-49.